CLINICAL TRIAL: NCT03619824
Title: Neoadjuvant Sintilimab (PD-1 Antibody)-Chemotherapy and Concurrent Sintilimab-chemoradiation in Locoregionally-advanced Nasopharyngeal Carcinoma: a Single-arm, Phase 2 Clinical Trial
Brief Title: PD-1 Blockade Combined With Definitive Chemoradiation in Locoregionally-advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-090-01
Record Dates: First submitted 2018-07-30; First posted 2018-08-08 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — sintilimab; spartalizumab; Gemcitabine; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 66-70Gy will be given in six to seven weeks. Concurrent cisplatin 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT. Sintilimab 200mg will be given every 3 weeks for 6 cycles, started on day 1 of induction chemotherapy.
  Interventions: Drug: Sintilimab; Drug: Gemcitabine; Drug: Cisplatin; Radiation: intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg ivdrip, every 3 weeks for 6 cycles
  Other Names: IBI308; PD-1 antibody
Drug: Gemcitabine — Gemcitabine 1g/m2, d1 & 8 of every cycle, every 3 weeks for 3 cycles before radiation.
Drug: Cisplatin — Induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiation Concurrent cisplatin 100mg/m2, every 3 weeks for 2 cycles during radiation
  Other Names: DDP
Radiation: intensity-modulated radiotherapy — Definitive IMRT of 66-70Gy will be given in six to seven weeks.
  Other Names: IMRT

SUMMARY:
This trial plans to enroll 40 patients with stage III-IVA (AJCC 8th, except T3N0-1 or T4N0) locoregionally-advanced nasopharyngeal carcinoma (NPC). Patients will receive 3 cycles of induction chemotherapy with gemcitabine and cisplatin and concurrent cisplatin-radiation. All patients will receive intensity-modulated radiotherapy (IMRT). Sintilimab will begin on day 1 of induction chemotherapy and continue every 3 weeks for 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed nasopharyngeal carcinoma.
2. Tumor staged as III-IVA (AJCC 8th, except T3N0-1 or T4N0).
3. ECOG performance status ≤1.
4. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.
5. Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN.
6. Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).
7. Patients must be informed of the investigational nature of this study and give written informed consent.
8. Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug.

Exclusion Criteria:

1. Age > 65 or < 18.
2. Hepatitis B surface antigen (HBsAg) positive and HBV DNA >1×10e3 copies/ml
3. Hepatitis C virus (HCV) antibody positive
4. Has active autoimmune disease, except type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
5. Has a known history of interstitial lung disease.
6. Has any condition that required systemic corticosteroid (equivalent to prednisone >10mg/d) or other immunosuppressive therapy within 28 days before informed consent. Patients received systemic corticosteroid equivalent to prednisone ≤10mg/d, inhale or topical corticosteroid will be allowed.
7. Has received a live vaccine within 30 days before informed consent or will receive a live vaccine in the near future.
8. Is pregnant or breastfeeding.
9. Prior malignancy within 5 years, except in situ cancer, adequately treated non-melanoma skin cancer, and papillary thyroid carcinoma.
10. Has known allergy to large molecule protein products or any compound of sintilimab.
11. Has a known history of human immunodeficiency virus (HIV) infection.
12. Any other condition, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic therapy, mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Immune-related adverse events (irAEs) and serious adverse events (irSAEs) | From the date of informed consent to 100 days after treatment
  Graded according to CTCAE V5.0
All adverse events (AEs) and serious adverse events (SAEs) | From the date of informed consent to 100 days after treatment
  Graded according to CTCAE V5.0

SECONDARY OUTCOMES:
The proportion of patients who completed radiation within 8 weeks | 8 weeks
The proportion of patients who completed 6 cycles of sintilimab | From the date of informed consent to the end of treatment, assessed up to 20 weeks.
Failure-free survival | 3 years
  calculated from the date of informed consent to the date of locoregional failure, distant failure, or death from any cause, whichever occurred first.
Overall survival | 3 years
  calculated from the date of informed consent to the date of death from any cause.
Distant failure-free survival | 3 years
  calculated from the date of informed consent to the date of distant metastasis.
Locoregional failure-free survival | 3 years
  calculated from the date of informed consent to the the date of locoregional persistence or 1st locoregional recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, Principal Investigator — Sun Yat-sen University
Locations (1):
- SUN YAT-SEN UNIVERSITY cANCER CENTER, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li XM, Zhang XM, Li JY, Jiang N, Chen L, Tang LL, Mao YP, Li WF, Zhou GQ, Li YQ, Liu N, Zhang Y, Ma J. The immune modulation effects of gemcitabine plus cisplatin induction chemotherapy in nasopharyngeal carcinoma. Cancer Med. 2022 Sep;11(18):3437-3444. doi: 10.1002/cam4.4705. Epub 2022 Mar 30. PMID 35355438